CLINICAL TRIAL: NCT04867941
Title: A 2-Part, Open-Label, Single-Dose Study to Investigate the Influence of Hepatic Insufficiency on the Pharmacokinetics of ACP-196
Brief Title: A Study to Evaluate the Effect of Hepatic Insufficiency on the Pharmacokinetics (PK) of ACP-196
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-HI-001
Record Dates: First submitted 2021-04-28; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Hepatic Insufficiency
Keywords: ACP-196; Healthy participants; Mild hepatic impairment; Moderate hepatic impairment; Severe hepatic impairment; Pharmacokinetics; PK; Safety
MeSH Terms: conditions — Hepatic Insufficiency | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part1: Mild hepatic insufficiency (Experimental): Participants with mild hepatic insufficiency will receive a single oral dose of 50 mg ACP-196 (2 x 25 mg capsules) on Day 1 of the study.
  Interventions: Drug: ACP-196
- Part 1: Moderate hepatic insufficiency (Experimental): Participants with moderate hepatic insufficiency will receive a single oral dose of 50 mg ACP-196 (2 x 25 mg capsules) on Day 1 of the study.
  Interventions: Drug: ACP-196
- Part 1: Normal hepatic function (Experimental): Participants with normal hepatic function will receive a single oral dose of 50 mgACP-196 (2 x 25 mg capsules) on Day 1 of the study.
  Interventions: Drug: ACP-196
- Part 2: Severe hepatic insufficiency (Experimental): Participants with sever hepatic insufficiency will receive a single oral dose of 50 mg ACP-196 (2 x 25 mg capsules) on Day 1 of the study.
  Interventions: Drug: ACP-196

INTERVENTIONS:
Drug: ACP-196 — All study participants will receive a single oral dose of 50 mg ACP-196 (2 x 25 mg capsules) on Day 1 of the study.
  Other Names: Acalabrutinib

SUMMARY:
The study will evaluate the influence of hepatic insufficiency on the PK of ACP-196.

DETAILED DESCRIPTION:
This is a 2-part study. Part 1 of the study will compare the PK of ACP-196 in participants with mild hepatic insufficiency (a score of 5 to 6, on the Child-Pugh scale) and moderate hepatic insufficiency (a score of 7 to 9, on the Child-Pugh scale) to healthy (mean) matched control participants for age and weight. Part 2 of the study, if it is conducted, will compare the PK of ACP-196 in participants with severe hepatic insufficiency (a score of 10 to 15 on the Child-Pugh scale) to the healthy control participants from Part 1. In Part 1, 6 participants with mild hepatic insufficiency, 6 participants with moderate hepatic, and 6 healthy control participants matched to the hepatic insufficiency groups according to mean age and mean weight will be enrolled. In Part 2, if conducted, 6 participants with severe hepatic insufficiency will be enrolled. The control group of Part 1 will be used for Part 2 PK comparison. Participants will be screened within 28 days before the dose. Participants will be contacted approximately 14 days after the last dose of study drug administration to determine if any adverse event has occurred since the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Continuous non-smokers or smokers (of fewer than 20 cigarettes/day or the equivalent). Participants must agree to consume no more than 10 cigarettes or equivalent/day from 24 hours before dosing and throughout the period of sample collection.
* Women participants must be of non-child bearing status and must have negative serum pregnancy test.
* Men of reproductible potential must be willing to abstain from heterosexual intercourse or refrain from sperm donation or use contraception during the study and through 90 days after the last dose of study drug.

Hepatic impaired participants:

* Body mass index (BMI) >= 19 and <= 40 kg/m^2, at screening.
* Have medical history, physical examination, vital signs, 12-lead ECGs, and laboratory safety tests consistent with a diagnosis of hepatic impairment, but is otherwise judged to be in good health as determined by the principal investigator (PI).
* Participant has a diagnosis of chronic (> 6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) hepatic insufficiency with features of cirrhosis due to any etiology.
* Part 1 only: Mild - Participant's score on the Child-Pugh scale must range from 5 to 6 (mild hepatic insufficiency) at screening. Moderate - Participant's score on the Child-Pugh scale must range from 7 to 9 (moderate hepatic insufficiency) at screening. For participants who have compensated hepatic insufficiency while on medical therapy, they should be classified by their pretreatment parameters.
* Part 2 only: Severe - Participant's score on the Child-Pugh scale must range from 10 to 15 (severe hepatic insufficiency) at screening. For participant's who have compensated hepatic insufficiency while on medical therapy, they should be classified by their pretreatment parameters.

Healthy control participants only:

* BMI >= 19 and <= 40 kg/m^2 at screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECGs, as deemed by the PI. Liver function tests, and serum bilirubin, must be <= the upper limit of normal at screening.

Exclusion Criteria:

All participants:

* History or presence of clinically significant or unstable medical or psychiatric condition or disease in the opinion of the PI.
* Participant is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* Any clinically significant condition that may affect ACP-196 absorption in the opinion of the PI, including gastric restrictions and bariatric surgery (eg, gastric bypass).
* Unable to refrain from or anticipates use of medicines defined in the protocol..
* Have been on a diet incompatible with the on-study diet, in the opinion of the PI, within the 28 days before the dose of study drug, and throughout the study.

Hepatic impaired participants only:

* History or presence of drug abuse within the past 2 years before screening.
* Positive results for the urine or breathalyzer alcohol test and/or urine drug screen at screening or check-in, unless the positive drug screen is due to prescription drug use and is approved by the PI and Acerta Pharma's medical monitor.
* Known history of HIV or hepatitis B virus (HBV) or active infection with hepatitis C virus (HCV). During screening, participants who have active HCV infection or unstable levels of transaminase consistent with active Hepatitis C, will be excluded.
* No hepatic impaired participant will be dosed in both Part 1 and Part 2.

Healthy control participants only:

* History or presence of clinically significant thyroid disease, in the opinion of the PI.
* History or presence of alcoholism and/or drug abuse within the past 2 years before screening.
* Positive results for the urine or breathalyzer alcohol test and/or urine drug screen at screening.
* Positive results at screening for hepatitis B surface antigen or HCV.
* Seated blood pressure is less than 90/40 mmHg or greater than 150/95 mmHg at screening.
* Seated heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at screening.
* Hemoglobin level below the lower limit of normal at screening, and considered clinically significant by the PI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10-21 (Actual); Primary Completion 2015-02-02 (Actual); Study Completion 2015-02-02 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of ACP-196 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours (hrs) for all arms, additional timepoints at 36 and 48 hrs post dose for mild/moderate/severe hepatic insufficiency arms
Maximum Observed Plasma Concentration (Cmax) of ACP-196 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours (hrs) for all arms, additional timepoints at 36 and 48 hrs post dose for mild/moderate/severe hepatic insufficiency arms

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time 0 To Time of Last Measurable Concentration (AUC0-last) of ACP-196 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours (hrs) for all arms, additional timepoints at 36 and 48 hrs post dose for mild/moderate/severe hepatic insufficiency arms
Area Under the Plasma Concentration-time Curve From Time 0 To 24 Hours (AUC0-24) of ACP-196 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours (hrs) for all arms, additional timepoints at 36 and 48 hrs post dose for mild/moderate/severe hepatic insufficiency arms
Percent of AUC0inf Extrapolated (AUC%extrap) of ACP-196 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours (hrs) for all arms, additional timepoints at 36 and 48 hrs post dose for mild/moderate/severe hepatic insufficiency arms
Time of the Maximum Measured Plasma Concentration (Tmax) of ACP-196 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours (hrs) for all arms, additional timepoints at 36 and 48 hrs post dose for mild/moderate/severe hepatic insufficiency arms
Time of the Last Measurable Plasma Concentration (Tlast) of ACP-196 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours (hrs) for all arms, additional timepoints at 36 and 48 hrs post dose for mild/moderate/severe hepatic insufficiency arms
Apparent Terminal Elimination Rate Constant (λz) of ACP-196 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours (hrs) for all arms, additional timepoints at 36 and 48 hrs post dose for mild/moderate/severe hepatic insufficiency arms
Apparent Terminal Elimination Half-life (T1/2) of ACP-196 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours (hrs) for all arms, additional timepoints at 36 and 48 hrs post dose for mild/moderate/severe hepatic insufficiency arms
Apparent Total Body Clearance (CL/F) of ACP-196 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours (hrs) for all arms, additional timepoints at 36 and 48 hrs post dose for mild/moderate/severe hepatic insufficiency arms
Apparent Total Volume of Distribution (Vz/F) of ACP-196 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours (hrs) for all arms, additional timepoints at 36 and 48 hrs post dose for mild/moderate/severe hepatic insufficiency arms
Incidences of Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | From Day 1 through 14 days after the last dose (approximately 4 months)
Incidences of Abnormal Vital Signs and Physical Examinations Reported as TEAEs | Day 1 through Day 3
Incidences of Abnormal Electrocardiograms (ECGs) Reported as TEAEs | Day 1 through Day 3
Incidences of Abnormal Clinical Laboratory Parameters Reported as TEAEs | Day 1 through Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Priti Patel, MD, Study Director — Acerta Pharma BV
Locations (3):
- United States (3):
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home